CLINICAL TRIAL: NCT05909852
Title: A Randomized, Single-blind, Single-dose, 2-arm, Parallel-group Study to Determine the Pharmacokinetic Comparability of ABP 501 40 mg/0.4 mL (ABP 501-HCF) and ABP 501 40 mg/0.8 mL (ABP 501-LCF) in Healthy Adult Subjects
Brief Title: A Study Comparing the Pharmacokinetics (PK) of ABP 501 40 mg/0.4 mL (ABP 501-HCF) and ABP 501 40 mg/0.8 ml (ABP 501-LCF) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20200286
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Adalimumab
Keywords: Pharmacokinetics; Tumor necrosis factor; monoclonal antibody

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: ABP 501-HCF (Experimental): Participants will be administered a single SC dose of ABP 501-HCF on Day 1.
  Interventions: Drug: ABP 501-HCF
- Treatment B: ABP 501-LCF (Experimental): Participants will be administered a single SC dose of ABP 501-LCF on Day 1.
  Interventions: Drug: ABP 501-LCF

INTERVENTIONS:
Drug: ABP 501-HCF — Participants will receive a single-dose SC injection of ABP 501-HCF.
  Arms: Treatment A: ABP 501-HCF
Drug: ABP 501-LCF — Participants will receive a single-dose SC injection of ABP 501-LCF
  Arms: Treatment B: ABP 501-LCF

SUMMARY:
To determine the pharmacokinetic (PK) comparability of ABP 501 40 mg/0.4 mL (ABP 501-HCF) compared to ABP 501 40 mg/0.8 mL (ABP 501-LCF) following single-dose subcutaneous (SC) injection, as assessed principally by area under the serum concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf) and maximum observed serum concentration (Cmax) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed consent form (ICF) before any study-specific procedures are performed.
* Healthy adult male or female participants between 18 and 55 years of age, inclusive, at the time of screening.
* Body weight of ≥ 50 kg and ≤ 90 kg.
* Body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive. (BMI = weight [kg]/height[m^2]).
* Normal or clinically acceptable physical examination, clinical laboratory test values, vital signs, and 12-lead electrocardiogram as determined by the investigator, at screening and/or on Day -1. This determination must be recorded in the participant's source documents and initialed by the investigator.
* Chest X-ray with no evidence of current, active tuberculosis (TB) or previous (inactive) TB, other active infections, malignancy, or other clinically significant abnormalities, taken at screening or within 3 months prior to day 1 and read by a qualified radiologist. Chest X-ray may be substituted by a high resolution chest computed tomography (CT) or chest magnetic resonance imaging (MRI), if available within 3 months prior to screening.
* Participants must be able to communicate effectively with the study personnel.

Exclusion Criteria:

* Female participant who is pregnant or breastfeeding or planning to become pregnant while participating in the study and for at least 5 months after the last dose of study drug.
* Female of childbearing potential who is sexually active with male partner and is unwilling to use an effective method of birth control. Effective birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 5 months after the last dose of study drug. Females of childbearing potential must also agree not to donate eggs (ova, oocytes for the purpose of assisted reproduction) for at least 5 months after the last dose of study drug.
* Female participant of childbearing potential with a positive serum pregnancy test at screening or a positive urine pregnancy test on Day -1.
* History or evidence of a clinically significant condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion. Includes history of demyelinating disease or neurologic symptoms suggestive of demyelinating disease.
* History or presence of conditions or comorbidity known to interfere with the distribution, metabolism, or excretion of drugs or which may interfere with study assessment, including assessment of injection site, in the opinion of the investigator.
* Evidence of any bacterial, viral, parasitic, or systemic fungal infection within the past 30 days prior to randomization (e.g., upper respiratory tract infection, viral syndrome, flu-like symptoms).
* History or clinically significant chronic and/or recurrent infections, including but not limited to herpes zoster infection within 3 months prior to screening, renal or urinary tract infections (e.g., chronic pyelonephritis, recurrent cystitis), fungal infection (mucocutaneous candidiasis), or chronic pulmonary infection (e.g., bronchiectasis).
* Evidence of recent (within 3 months prior to randomization) infection requiring in-patient hospitalization or intravenous (IV) systemic anti-infectives.
* Participant has active TB, latent TB (defined as a positive result QuantiFERON® TB Gold test [or interferon gamma releasing assay {IGRA}] without any signs or symptoms of TB), a history of TB, or had close contact with a person with active TB within 12 weeks prior to administration of the study drug (Day 1); or participant has a repeat indeterminate QuantiFERON® TB Gold test (or IGRA equivalent).
* History of invasive systemic fungal infections (e.g., coccidiomycosis, histoplasmosis etc.) prior to or during the screening period.
* History of non-tuberculous mycobacterial or opportunistic infection 3 months prior to screening.
* History of surgery or major trauma within 3 months of screening, or surgery (requiring general anesthesia) planned during the study.
* History of malignancy of any type other than completely cured non-metastatic squamous or basal cell carcinoma of the skin, or in situ carcinoma of the uterine cervix within 5 years prior to screening.
* Positive screen for hepatitis B virus surface antigen, hepatitis B core antibody, or hepatitis C virus antibody.
* History of human immunodeficiency virus (HIV) or positive HIV serology at screening.
* Positive screen for alcohol and/or potential drugs of abuse (urine drug screen) at screening or prior to randomization or history of alcohol and/or substance abuse within the last 12 months prior to screening.
* Receiving or has received any investigational drug including investigational vaccine (or is currently using an investigational device) within the 30 days or 5 half-lives (whichever is longer) prior to randomization.
* Use of any over-the-counter or prescription medicines within the 14 days or 5 half-lives (whichever is longer) prior to randomization.
* Donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months prior to study drug administration.
* Received live viral or live bacterial vaccines within 3 months prior to randomization or is scheduled to receive a live vaccine within 3 months following treatment with study drug.
* Known or suspected intolerance, allergic reactions, or hypersensitivity to products derived from mammalian cells lines or any biologic medication.
* Known allergy to natural rubber (a derivative of latex).
* Previously received adalimumab or a biosimilar of adalimumab (investigational or marketed).
* Inability or unwillingness to reside at the clinical pharmacology unit for 2 consecutive days or inability to be available for follow-up assessments or protocol-required procedures.
* Participants who smoked >10 cigarettes per day within the last 3 months or not able to abide by the smoking policy of the site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 372 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
AUCinf of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Cmax of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63

SECONDARY OUTCOMES:
AUC from Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Time at which Cmax is Observed (Tmax) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Terminal Elimination Half-life (t1/2) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Apparent Clearance (CL/F) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Apparent Volume of Distribution (Vz/F) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Mean Residence Time (MRT) of ABP 501-HCF and ABP 501-LCF | Pre-dose (Day 1), 8 hours post-dose (Day 1), Days 2 to 9, Days 11, 14, 16, 22, 29, 36, 43, 50, 57, and 63
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Day 1 until Day 63
  An adverse event (AE) is an untoward medical occurrence in a clinical study irrespective of a causal relationship with the study treatment. The number of participants with TEAEs including serious AEs, clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests.
Number of Participants with an Event of Interest | Day 1 until Day 63
Number of Participants with Binding and Neutralizing Anti-drug Antibodies | Pre-dose Day 1, Day 16, Day 29, and Day 63

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - WCCT Global, Inc, Cypress, California
  - Qps-Mra, Llc, South Miami, Florida
  - Pharmaceutical Research Associates, Inc, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com